CLINICAL TRIAL: NCT04752865
Title: Effects of Cytotoxic Chemotherapy and PARP Inhibition on the Genomic Contexture of Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: TR_NACT_OV/17
Record Dates: First submitted 2020-12-17; First posted 2021-02-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissues will be histologically reviewed for tumor presence and evaluated for tumor cell content (TCC%) and adequacy for genotyping, tumor lymphocytic infiltrates (TILs) and further morphologic features (presence of intraepithelial lymphocytes, micro- and macro-necrosis, hemorrhagic infiltrates, specific and heterogeneous morphologic patterns) that will be recorded in detail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EFFECTS OF CYTOTOXIC CHEMOTHERAPY AND PARP INHIBITION ON THE GENOMIC CONTEXTURE OF OVARIAN CANCER: TR_NACT_OV/17 In order to approach the above open questions, ultimately aiming in understanding the effects of cancer drugs on tumor biology and hence in selecting the proper drugs for the patients in the context of Precision Medicine, the objective of this study is to study the genomic characteristics of ovarian tumors before and after treatment with classic neoadjuvant chemotherapy (NACT) and with the more recently approved PARP inhibitor olaparib.

ELIGIBILITY:
Inclusion Criteria:

* ovarian cancer eligible for neoadjuvant chemotherapy

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with ovarian cancer eligible for neoadjuvant chemotherapy. The investigators examined changes in tissue molecular profile. The investigators examine tissue molecular profile at diagnosis and after the end of neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
assesment of genomic characteristics of ovarian tumors at the diagnosis | 4 years
assesment of genomic characteristics of ovarian tumors after treatment with neoadjuvant platinum-based chemotherapy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Adamantia Nikolaidi, Study Chair — HECOG
Locations (1):
- Adamantia Nikolaidi, Athens, Greece